CLINICAL TRIAL: NCT01519024
Title: Poorer Postural Control in Women With Breast Hypertrophy.
Brief Title: Postural Control in Breast Hypertrophy
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FRACINI_1
Record Dates: First submitted 2012-01-23; First posted 2012-01-26 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Hypertrophy; Sensation Disorders
Keywords: hypertrophy; breast; postural balance
MeSH Terms: conditions — Hypertrophy; Sensation Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Women with breast hypertrophy: Fourteen women with breast hypertrophy
- Women without breast hypertrophy.: Fourteen women without breast hypertrophy for de control group (CG).

SUMMARY:
Principles of motor control suggest that breast hypertrophy can lead to sensoriomotor alterations and impairment in body balance due to postural misalignment. The investigators conducted this study to evaluate the postural control with different sensorial information condition in women with breast hypertrophy.

DETAILED DESCRIPTION:
Up to the moment, changes caused by breast hypertrophy are described based on the alteration of body mass distribution leading to an impact of psychological and physical aspects. However, the investigators hypothesize that due to alterations in postural alignment, sensoriomotor inputs are also impaired and postural or motor control are ultimately compromised.

ELIGIBILITY:
Inclusion Criteria:

* For the breast hypertrophy group, the women had to be in attendance in the Department of Plastic Surgery and Department of Gynecology of Clinical Hospital.

Exclusion Criteria:

* For both groups:

  * rheumatic, neurological, respiratory and vestibular conditions due to possible balance alterations

Ages: 24 Years to 73 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The fourteen women for breast hypertropy group were recruited from the Department of Plastic Surgery and Department of Gynecology of Clinical Hospital, Faculty of Medicine, University of São Paulo, and the fourteen women of control group (without breast hypertrophy)was compound by women dwelling community.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2010-04; Primary Completion 2011-02 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clarice Tanaka, PhD, Principal Investigator — Full Professor - Department of Physical Therapy, Communication Science & Disorders, Occupational Therapy, Faculty of Medicine - USP
Locations (1):
- Physical Therapy, Speech and Occupational Therapy Department, School of Medicine: University of São Paulo, São Paulo, São Paulo, Brazil